CLINICAL TRIAL: NCT01655888
Title: A SECOND-LINE, SINGLE ARM, PHASE II CLINICAL STUDY WITH TREMELIMUMAB, A FULLY HUMAN ANTI-CTLA-4 MONOCLONAL ANTIBODY, AS MONOTHERAPY IN PATIENTS WITH UNRESECTABLE MALIGNANT MESOTHELIOMA. The MESOT-TREM-2012
Brief Title: The Anti-CTLA-4 Monoclonal Antibody Tremelimumab in Malignant Mesothelioma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Universitaria Senese (Other)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Principal Investigator, Michele Maio, Head of Medical Oncology and Immunotherapy Unit, Azienda Ospedaliera Universitaria Senese
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MESOT-TREM-2012; 2012-002762-12 (EudraCT Number)
Record Dates: First submitted 2012-07-31; First posted 2012-08-02 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Malignant Mesothelioma
Keywords: Tremelimumab; anti-CTLA-4 monoclonal antibody; malignant mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm with Tremelimumab (Experimental): Tremelimumab: 10mg/Kg ev day 1 every 4 weeks for 6 doses in induction phase, then every 12 weeks in maintenance phase until disease progression of severe toxicity
  Interventions: Drug: Tremelimumab

INTERVENTIONS:
Drug: Tremelimumab — Tremelimumab is administered as endovenous infusion
  Other Names: CP-675,206

SUMMARY:
RATIONAL: Preliminary results fron the Study MESOT-TREM-2012 indicate a promising activity of tremelimumab in malignant mesothelioma (MM) patients.

PURPOSE: The proposed study MESOT-TREM-2012 aims to explore the efficacy of a more intensive schedule of treatment with tremelimumab in 29 MM patients. Subjects will receive investigational product every 4 weeks (wks) for 6 doses, followed by doses every 12 wks until confirmed disease progression.

DETAILED DESCRIPTION:
Primary endpoint:

1) To assess the rate of objective clinical complete response (CR) or partial response (PR)

Secondary endpoints:

1. To define toxicity profile according to NCI CT-CAE V. 3
2. To assess the overall survival (OS)
3. To estimate disease control rate (DCR) (proportion of patients with best response of CR+PR+SD) according to the modified Recist criteria
4. To assess the progression-free survival in treated patients according to modified Recist criteria
5. To evaluate qualitative and quantitative changes in cellular and humoral immune responses

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed MM
* Have received only one prior systemic chemotherapy platinum-based regimen for advanced MM
* Measurable disease, defined at least 1 unidimensionally measurable lesion > 20 mm by conventional techniques or > 10 mm by spiral CT scan (modified RECIST criteria)
* Disease not amenable to curative surgery
* No known brain metastasis
* Age 18 and over
* Performance status 0-2
* Life expectancy > 12 weeks
* Adequate hematologic, hepatic and renal function
* Platelet count > 75000/mm3
* Absolute granulocyte count > 1000/mm3
* Hemoglobin > 9 g/dL
* Bilirubin total < 1.5 x ULN (Upper limited normal), except patients with documented Gilbert's syndrome, who must have a total bilirubin < 3.0 mg/dl
* AST and ALT < 2.5 x ULN ( < 5 x ULN if documented liver metastasis are present)
* Creatinine level < 2mg/dl or calculated creatinine clearance > 60 mL/min as determined by the Cockcroft Gault equation.
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Patient must be willing and able to provide written informed consent, and the trial have to be approved by the institutional review board at each institution

Exclusion Criteria:

* Symptomatic chronic inflammatory or autoimmune disease
* Active hepatitis B or C
* Prior treatment with tremelimumab or other anti-CTLA-4 antibody or anti-PD1, anti-PDL-1 agents
* Clinically relevant cardiovascular disease
* History of psychiatric disabilities, potentially interfering with the capability of giving adequate informed consent
* Uncontrolled active infections
* Other concurrent chemotherapy, immunotherapy, radiotherapy or investigational agents
* History of other malignancies except for adequately treated basal cell carcinoma or squamous cell skin cancer or carcinoma of cervix, unless the patient has been disease-free for at least 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
To determine the objective response | Weeks 24
  The objective response is defined as a confirmed complete response (CR), or partial response (PR) according to the modified RECIST Criteria for pleural mesothelioma and the immune-related (ir) Response Criteria

SECONDARY OUTCOMES:
Disease control rate (DCR) | 1 year
  DCR is the proportion of treated subjects that achieved confirmed CR or PR or stable disease (SD) The DCR is assessed using the modified RECIST Criteria for pleural mesothelioma umor assessment and the the immune-related response criteria
Safety | 3 years
  The assessment of safety includes serious and non-serious adverse events according to NCI-CTC criteria version 3.0. In addition, laboratory evaluation, abnormal vital signs and physycal examination findings are also included.
Progression free survival | 1 years
  Progression free survival is computed from the first day of study treatment to the day of documented progression according to the modified RECIST Criteria for pleural mesothelioma or death, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Michele Maio, MD, Principal Investigator — Medical Oncology and Immunotherapy Unit, University Hospital of Siena, Italy; Luana Calabrò, MD, Principal Investigator — Medical Oncology and Immunotherapy, University Hospital of Siena, Italy
Locations (1):
- Medical Oncology and Immunotherapy Unit, University Hospital of Siena, Siena, Italy

REFERENCES:
- [Derived] Calabro L, Morra A, Fonsatti E, Cutaia O, Fazio C, Annesi D, Lenoci M, Amato G, Danielli R, Altomonte M, Giannarelli D, Di Giacomo AM, Maio M. Efficacy and safety of an intensified schedule of tremelimumab for chemotherapy-resistant malignant mesothelioma: an open-label, single-arm, phase 2 study. Lancet Respir Med. 2015 Apr;3(4):301-9. doi: 10.1016/S2213-2600(15)00092-2. Epub 2015 Mar 26. PMID 25819643